CLINICAL TRIAL: NCT04809896
Title: Homemade Fenestrated Physician-modified Stent-grafts for Arch Aortic Degenerative Aneurysm
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0161
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Aortic Arch Aneurysm
Keywords: Proximal descending aorta aneurism; Proximal and distal neck (length >20mm et diameter >20mm and <40mm; thoracic endovascular aortic repair; Intra-abdominal septic complications
MeSH Terms: conditions — Aneurysm, Aortic Arch

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim was to evaluate early and medium-term outcomes of single and double fenestrated physician-modified endovascular grafts (PMEGs) for endovascular aortic arch degenerative aneursym repair.

The evolution of stent-graft technology recently has meant the development of custom-made branched stent-grafts to achieve total endovascular aortic arch repair for high-risks patients. The disadvantages of custom-made include manufacture and deliver times for urgent cases and the associated high costs. Unfortunately there is also a high rate of embolization associated with this approach probably related to the complexity of deploying a multi-branched unibody stent-graft. A further alternative is physician modified endografts (PMEGs) for zone 0 TEVAR involving the deployment of a conventional stent-graft device ex-vivo, fashioning of customized fenestrations (for supra aortic trunk) and re-constrainment into the delivery system. The authors have previously shown the feasability in vitro and they have reported their experience for arch aortic lesion. The aim of this study is to evaluate the outcomes for aortic arch degenerative aneursym repair which is the most risky procedure

ELIGIBILITY:
Inclusion criteria:

- patients operated on in our department between 2000 and January 2020 for a thoracic endoprosthesis

Exclusion Criteria:

- Patient who reject the study protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population requiring this procedure is elderly, with major comorbidities and some of these indications are given in an emergency context.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Rate of retrograde aortic dissection | day 1
  Rate of retrograde aortic dissection

SECONDARY OUTCOMES:
Rate of endoleak | day 1
  Rate of endoleak
Rate of stroke | day 1
  Rate of stroke
Rate of Mortality | 30 days
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: ludovic CANAUD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC